CLINICAL TRIAL: NCT05460923
Title: Comparison of Pelvic Neuromuscular Facilitation and Swiss Ball Exercises on Trunk Control in Children With Diaplegic Cerebral Palsy
Brief Title: Pelvic Neuromuscular Facilitation and Swiss Ball Exercises on Trunk Control in Children With Diaplegic CP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0716
Record Dates: First submitted 2022-07-14; First posted 2022-07-15 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy, Trunk Control Training, Proprioceptive Neuromuscular Facilitation Approach, Swiss ball, Trunk Control Measurement Scale.
MeSH Terms: conditions — Cerebral Palsy | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Swiss Ball Exercises (Experimental): Swiss ball exercises along with baseline treatment trunk twists,
  Interventions: Other: Swiss Ball Exercises
- Proprioceptive Neuromuscular Facilitation (Experimental): pelvic neuromuscular facilitation techniques including various PNF movement patterns along with the baseline treatment
  Interventions: Other: Proprioceptive Neuromuscular Facilitation

INTERVENTIONS:
Other: Proprioceptive Neuromuscular Facilitation — including trunk twists, supine to sit, knee to chest, crawling, and bridges. Every session will be 45 minutes. Patients will be given 5 sessions per week and the study will last for 12 months
  Arms: Proprioceptive Neuromuscular Facilitation
Other: Swiss Ball Exercises — trunk twists, supine to sit, knee to chest, crawling, and bridges. Every session will be 45 minutes. Patients will be given 5 sessions per week and the study will last for 12 months
  Arms: Swiss Ball Exercises

SUMMARY:
Cerebral palsy is an umbrella term that covers a group of non-progressive motor impairment syndromes that are associated with abnormalities in the brain particularly during the early stages of its development. CP usually involves a number of musculoskeletal and neurological problems they include spasticity, contractures, dystonia, abnormal growth, poor trunk control, and poor balance. Poor trunk control leads to a disturbance in activities of daily living along with postural issues. PNF techniques and Swiss ball exercises target the trunk muscles by stimulating the proprioceptors and by allowing maximum resistance to them respectively. The aim of the study is to do a comparison of Pelvic neuromuscular facilitation techniques and Swiss ball exercises in improving trunk control in children with diplegic cerebral palsy.

DETAILED DESCRIPTION:
The studies conducted in the past were focused on finding out the effect of proprioceptive neuromuscular facilitation techniques on the lower extremities of children suffering from diplegic cerebral palsy. The effects of PNF on trunk control the children suffering from diplegic CP are nearly minimal. In addition to PNF, the literature shows that studies have been conducted to find the effects of Swiss ball training exercise on trunk control of the post-stroke patients however there is very little research on the effects of Swiss ball training in children suffering from diplegic CP. Even if the studies are conducted the time duration of the studies are not enough to gain the maximum outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with no trunk control
* Age between 5-12 years
* Patients with diplegia

Exclusion Criteria:

* Patients with Cognitive impairment
* Patients with comorbidities
* Patients who are unable to follow instructions

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2022-09-25 (Estimated); Study Completion 2022-11-28 (Estimated)

PRIMARY OUTCOMES:
Trunk Control Measurement Scale | 8th week
  The Trunk Control Measurement Scale is a clinical tool that is used in order to measure the trunk control. The scale is used in the areas of assessment of non-vestibular balance and functional mobility
GMFC | 8th week
  The Gross Motor Function Classification System or GMFCS is a 5 level clinical classification system that describes the gross motor function of people with cerebral palsy on the basis of self-initiated movement abilities.

CONTACTS AND LOCATIONS:
Overall Officials: Wajiha Shahid, PhD, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - International Therapy Services Center, Lahore, Punjab Province
  - Rising Sun Institute, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No